CLINICAL TRIAL: NCT00886314
Title: Clown Doctors and a Sedative Premedicant for Children Undergoing Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Yaacov Gozal, MD, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 12345
Record Dates: First submitted 2009-02-17; First posted 2009-04-22 (Estimated); Last update posted 2009-10-20 (Estimated); Status verified 2009-02

CONDITIONS: Insomnia
Keywords: children; surgery; anxiety
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders | interventions — Midazolam

ARMS (2):
- midazolam (Active Comparator)
  Interventions: Drug: midazolam
- clown doctor (Active Comparator)
  Interventions: Other: clown doctor

INTERVENTIONS:
Drug: midazolam — Children in this group will be premedicated with oral midazolam syrup (0.3 mg.kg) at least 15 minutes before the surgical procedure and one of the parents will be present throughout the anesthesia induction process.
  Arms: midazolam
Other: clown doctor — Children will interact with clowns before entering the operating room and will stay with them and one of the parents throughout the anesthesia induction process.
  Arms: clown doctor

SUMMARY:
The purpose of the present investigation will be to determine whether a combination of clown doctor and parental presence is more effective than a combination of sedative premedication and parental presence for reducing anxiety in children and their parents and for improving parental satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* children aged 2 to 12 yr, scheduled for minor surgery under general anesthesia will be included in the present study.

Exclusion Criteria:

* Children with prematurity, development delay, previous anesthetic experience will be excluded from this study

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2009-06; Primary Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Preoperative anxiety | Prior to induction of anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Yaacov Gozal, MD, Principal Investigator — Shaare Zedek Medical Center, Jerusalem, Israel
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel